CLINICAL TRIAL: NCT07245030
Title: A Comparative Evaluation of the Effectiveness of Virtual Reality Eyewear vs Show-Do Technique on Dental Anxiety and Behavior in a Group of Children With Different Levels of Hearing Impairment During Dental Prophylaxis Procedure: A Randomized Controlled Trial
Brief Title: Effectiveness of Virtual Reality vs Show-Do Technique on Dental Anxiety in Children With Hearing Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Principal Investigator, Tamara Saleh, general practitioner, October University for Modern Sciences and Arts
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Tamara MSA University
Record Dates: First submitted 2025-11-16; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Dental Anxiety of Hearing Impairment
Keywords: dental prophylaxis procedure; scaling; polishing; oral hygiene instructions; virtual reality; Anxiety; behavioral; hearing impairment
MeSH Terms: conditions — Anxiety Disorders; Behavior; Hearing Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children with different levels of hearing impairment, using Show-Do Technique in combined with VR ey (Experimental): A- Show-Do Technique:
  Description: This technique will be integrated with the VR eyewear intervention to enhance understanding and comfort. The show-do technique involves:
  * Show: The child will be shown the dental tools and explain their purpose, possibly using visual aids or models.
  * Do: The procedure will be Performed as explained with continuous reassurance and support.
  B- Virtual Reality Component:
  Participants in this group will experience a virtual reality (VR) eyewear in an environment designed to distract them during dental prophylaxis procedure. The VR content will be age-appropriate and engaging, and featuring interactive (e.g., Fun animations, and Cartoons).
  Implementation:
  Before the dental treatment and after the implementation with show-do, children will be fitted with VR eyewear, where the aim is to immerse the child in the VR experience to reduce their focus on the dental treatment.
  Duration:
  • The VR eyewear experience will last for the duration of t
  Interventions: Device: virtual reality distraction
- Children with different levels of hearing impairment, using Show-Do Technique: (Active Comparator): Participants in this group will receive the standard show-do technique without the VR eyewear distraction. The same steps (Show, Do) will be employed to prepare the child for the dental procedure, but without the use of VR technology.
  Interventions: Behavioral: show-do technique

INTERVENTIONS:
Device: virtual reality distraction — children wear virtual reality glasses during dental prophylaxis procedure to reduce dental anxiety and enhance patient's behavior.
  Arms: Children with different levels of hearing impairment, using Show-Do Technique in combined with VR ey
Behavioral: show-do technique — conventional behavioral technique where the dentist shows and then perform the procedure to reduce anxiety and build cooperation.
  Arms: Children with different levels of hearing impairment, using Show-Do Technique:

SUMMARY:
This randomized controlled clinical trial aims to compare the effectiveness of virtual reality (VR) eyewear used as a distraction method in combination with the Show-Do (SD) technique versus the traditional Show-Do technique alone in managing dental anxiety and improving behavioral responses among Egyptian children with different levels of hearing impairment during a dental prophylaxis procedure. The study will evaluate dental anxiety using pulse rate and the PJS-Pictorial Scale, while behavior will be assessed using the Frankl Behavior Rating Scale. The trial seeks to provide evidence-based guidance on the implementation of VR technology as an adjunctive non-pharmacological tool for children with communication barriers in pediatric dentistry.

DETAILED DESCRIPTION:
Dental anxiety is a common barrier to effective dental care in pediatric patients, particularly in children with special health care needs such as hearing impairment. Communication limitations can increase anxiety and reduce cooperation, complicating dental treatment delivery. Traditional non-pharmacological techniques such as the Show-Do (SD) method are widely used to reduce anxiety by familiarizing children with dental procedures through demonstration and gradual exposure. However, their effectiveness may be limited in children with hearing impairments, who may not fully understand auditory or verbal explanations.

Virtual reality (VR) eyewear represents an innovative behavioral management tool that immerses the child in an interactive and engaging virtual environment, thereby diverting attention away from the dental procedure and reducing anxiety. Evidence from recent systematic reviews indicates that VR interventions can significantly decrease pain perception and anxiety in pediatric medical and dental settings, yet studies specifically targeting children with hearing impairment remain scarce.

This randomized controlled trial will be conducted at the Pediatric Dentistry Department, Faculty of Dentistry, MSA University. Participants will include children with varying levels of hearing impairment requiring dental prophylaxis. Eligible participants will be randomly assigned in a 1:1 ratio to either the control group (Show-Do technique only) or the intervention group (Show-Do technique combined with VR eyewear). Dental anxiety will be measured objectively using pulse oximetry and subjectively using the PJS-Pictorial Scale, while behavior will be assessed using the Frankl Behavior Rating Scale.

The study is designed to generate clinical evidence regarding the efficacy of integrating VR eyewear with conventional behavioral management methods for children with communication challenges. The results are expected to contribute to the development of inclusive, non-pharmacological strategies to manage dental anxiety and improve cooperation among pediatric patients with hearing impairments, ultimately enhancing patient-centered care in pediatric dentistry.

ELIGIBILITY:
Inclusion Criteria:

1. Children with moderate to severe Hearing impairment.
2. Children require dental prophylaxis.
3. Apparently, Health Children.

Exclusion Criteria:

1. Children with severe cognitive impairment or developmental disorders.
2. Children who are unable or unwilling to cooperate with the study protocol or assessment.
3. Children with complicated systemic diseases.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
anxiety level (objective) | baseline (5 minutes before session), during treatment (real-time), and immediately post-treatment (within 5 minutes)
  tool: pulse oximeter unit: beats per minute

SECONDARY OUTCOMES:
anxiety level (subjective) | immediately before treatment (baseline), during treatment (real-time), and immediately after treatment (post-procedure)
  tool: Pictorial Judgement Scale for Anxiety Assessment (PJS-pictorial scale) unit: score 1-5, (1: means very happy, 5: means very anxious.)
behavior assessment | immediately before treatment (baseline), during treatment (real-time), and immediately after treatment (post-procedure)
  tool: Frankel rating scale unit: score 1-4 (1: means definitely negative and 4: means definitely positive)

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - October University for Modern Sciences and Arts, Giza, Giza Governorate
  - October University for Modern Sciences and Arts, Giza

IPD SHARING:
Plan to Share IPD: Yes